CLINICAL TRIAL: NCT04792359
Title: Intra and Inter- Observer Reproducibility of Ankle Dorsiflexion Measure With a New Tool
Acronym: EQUINOM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-A03518-31
Record Dates: First submitted 2021-03-04; First posted 2021-03-10 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Orthopedic
Keywords: Ankle-Dorsiflexion-Reproducibility -Measure-Orthopedic

STUDY DESIGN:
Intervention Model Description: Exploratory, interventional, prospective, uncontrolled, single arm, monocentric study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Equinometer (Experimental): Measurement with Equinometer
  Interventions: Device: Equinometer

INTERVENTIONS:
Device: Equinometer — Measurement of dorsiflexion of the ankle will be reproduced three times on each ankle in two positions, with a force applied

SUMMARY:
The Achilles' tendon is the largest and most resistant tendon in the body. When the triceps contracts, the Achilles' tendon is responsible for plantar flexion of the ankle. When the triceps are not contracted, the Achilles tendon is the main component in limiting dorsiflexion of the ankle, a major component of the gait pattern. The limitation of this dorsiflexion of the ankle can be caused by a shortening of the Achilles tendon.

This equine whose prevalence in the general population is greater than 50% according to Kowalski, appears to be a risk factor in many pathologies of the foot and ankle.

Currently, in clinical practice, the measurement of passive dorsiflexion of the ankle is empirically measured by the Silfverskiold test. However, the definition of a retraction varies according to the authors, in particular because of the absence of normalization of the force applied on the forefoot, or of the absence of uniformization of the angulation applied. This research is based on the hypothesis that a new measurement tool would be more efficient and more reproducible for measuring dorsiflexion of the ankle.

DETAILED DESCRIPTION:
The study includes the measure of dorsiflexion of the ankle with a new tool on volunteers. The measurement will be reproduced three times on each ankle in two positions, with a force applied by three different persons. The measurement will be automatically recorded then analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman, aged 18 years and more
* Student at the IFMK school (Paris)
* Participant without any trauma at the Achilles' tendon
* Participant who has been given appropriate information about the study objectives and who has given his/her express written and informed consent prior to conduct any study-related procedures.

Exclusion Criteria:

* Participant with a traumatic history of one of the two Achilles tendons
* Participant whose physical and / or psychological health is severely impaired, which according to the investigator may affect the participant's compliance with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2021-09-10 (Estimated); Study Completion 2021-09-10 (Estimated)

PRIMARY OUTCOMES:
Repeted measures of passive dorsiflexion of ankle using an equinometer at day1 | Day1 (single visit)
  measure defined by the angulation / force couple (degree / newton) in two positions of knee with three forces applied by three different persons using an equinometer including a dynanometer and a goniometer (both measurement automatically registred during the movement) at Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Julien BELDAME, MD, Principal Investigator — RGDS-Clinique Blomet
Locations (1):
- Clinique Blomet, Paris, France

IPD SHARING:
Plan to Share IPD: No